CLINICAL TRIAL: NCT05218005
Title: The Advancing Cardiac Care Unit-based Rapid Assessment and Treatment of hypErcholesterolemia (ACCURATE) Study
Brief Title: Advancing Cardiac Care Unit-based Rapid Assessment and Treatment of hypErcholesterolemia
Acronym: ACCURATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Genome British Columbia (Industry); Vancouver Coastal Health Research Institute (Other)
Responsible Party: Principal Investigator, Liam Brunham, Associate Professor, University of British Columbia
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: H21-00116
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Familial Hypercholesterolemia; Familial Hypercholesterolemia Due to Genetic Defect of Apolipoprotein B; Familial Hypercholesterolemia Due to Heterozygous LDL Receptor Mutation; Familial Hypercholesterolemia - Heterozygous; Acute Coronary Syndrome; NSTEMI - Non-ST Segment Elevation MI; STEMI; Familial Hypercholesterolemia With Hyperlipemia
Keywords: Familial hypercholesterolemia; hyperlipoproteinemia Type II; hyperlipoproteinemia type 2; familial hypercholesterolaemia; myocardial infarction; acute coronary syndrome; ST-elevated myocardial infarction; STEMI; non-ST-elevation myocardial infarction; NSTEMI; heart attack; genetic investigation; genetic testing; proprotein convertase subtilisin kexin 9; PCSK9; low-density lipoprotein receptor; LDLR; apolipoprotein B; APOB; low-density lipoprotein cholesterol; LDL-C
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction; Hyperlipoproteinemia Type III; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Two sequential groups of patients will be recruited. The first cohort will consist of a control group of patients presenting with acute coronary syndrome who will be treated according to usual standard-of-care. The second cohort will consist of patients presenting with acute coronary syndrome in whom research-based genetic testing for FH will be performed during hospitalization and the results returned to the treating physicians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation (No Intervention): Those admitted in the first 6 months of the study that meet the inclusion criteria. Patients will be treated according to the normal standard of care for acute coronary syndrome.
- Active-testing (Experimental): Those admitted between 6-18 months of the study meeting the inclusion criteria. Saliva samples will be collected for DNA testing.
  Interventions: Diagnostic Test: Research-based genetic test for Familial Hypercholesterolemia

INTERVENTIONS:
Diagnostic Test: Research-based genetic test for Familial Hypercholesterolemia — Next-generation targeted sequencing assay to identify DNA variants in genes known to cause Familial Hypercholesterolemia
  Arms: Active-testing

SUMMARY:
ACCURATE will test the hypothesis that opportunistic genetic testing for Familial Hypercholesterolemia (FH) in patients admitted to hospital with an acute coronary syndrome will increase the diagnosis of FH and will impact patient care and outcomes. The study will recruit patients admitted to hospital with an acute coronary syndrome, and research-based genetic testing will be conducted for known FH-causing genetic variants. The results will be returned to the patients' treating physicians. The primary endpoint will be the number of patients with a new diagnosis of FH. The secondary endpoints will be the proportion of patients who undergo intensification of lipid-lowering therapy, the lowest LDL cholesterol level achieved, and the proportion of patients reaching guideline recommended lipid targets in the 12 months after the index acute coronary syndrome.

DETAILED DESCRIPTION:
Familial hypercholesterolemia (FH) is an inherited condition characterized by elevated low-density lipoprotein cholesterol (LDL-C) levels and premature atherosclerotic cardiovascular disease (ASCVD). Despite being the most common inherited cardiovascular disorder, it is still highly underdiagnosed and undertreated worldwide. The Advancing Cardiac Care Unit-based Rapid Assessment and Treatment of hypErcholesterolemia (ACCURATE) study was designed to test the hypothesis that opportunistic genetic testing for FH among patients hospitalized for acute coronary syndrome (ACS) will increase the diagnosis of FH and improve patient outcomes. ACCURATE is a non-randomized, controlled trial of patients <60 years old admitted to an acute cardiac unit with ACS and elevated LDL-C levels. The first cohort will consist of a control group of patients presenting with ACS who will be treated according to usual standard-of-care. The second cohort will consist of patients presenting with ACS in whom research-based genetic testing for FH will be performed during hospitalization and the results returned to the treating physicians. The primary endpoint will be the number of patients with a new diagnosis of FH. The secondary endpoints will be the proportion of patients who undergo intensification of lipid-lowering therapy, the lowest LDL-C level achieved, and the proportion of patients reaching guideline recommended lipid targets in the 12 months after the index ACS. ACCURATE represents the first clinical trial of genetic testing for FH in the acute cardiac care setting and is expected to help identify optimal approaches to increase the diagnosis and treatment of FH.

ELIGIBILITY:
1. Age <60 years

   AND
2. Admitted to an acute cardiac unit with either:

   * A ST elevation myocardial infarction (STEMI), or
   * A non-ST elevation myocardial infarction (NSTEMI)

   AND
3. Maximum lipid level at the time of admission or during the prior 1 year of

   * LDL level ≥4 mmol/L (154 mg/dL) if not on a statin, or
   * LDL-C level ≥2.5 mmol/L (96 mg/dL) if on a statin prior to presentation, or
   * Non-HDL-C ≥4.6 mmol/L (177 mg/dL) if LDL-C not available

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a new diagnosis of FH | 1 year

SECONDARY OUTCOMES:
Proportion of patients in whom lipid-lowering medication intensified, as defined by an increase the dose of statin, or the addition of a non-statin lipid-lowering medication, in the first year after ACS | 1 year
Lowest LDL-cholesterol (LDL-C) level achieved in the first year after ACS | 1 year
Proportion of patients who achieve guideline recommended lipid targets in the first year after ACS | 1 year
  1. Canadian Cardiovascular Society Guidelines: LDL-C <1.8 mmol/L
  2. European Society of Cardiology Guidelines: ≥50% LDL-C reduction from baseline and LDL-C <1.4 mmol/L

OTHER OUTCOMES:
Rate of recurrent cardiovascular event in the first year after ACS | 1 year
  1. Unstable angina
  2. Myocardial infarction
  3. Urgent coronary revascularization
  4. Death

CONTACTS AND LOCATIONS:
Overall Officials: Liam Brunham, MD PhD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St.Pauls Hospital, Vancouver, British Columbia